CLINICAL TRIAL: NCT01646489
Title: A Phase 1, Open-Label, Drug Interaction Study to Assess Safety, Tolerability, and Pharmacokinetics of Co-Administered Miravirsen and Telaprevir in Healthy Subjects
Brief Title: Drug Interaction Study to Assess the Effect of Co-Administered Miravirsen and Telaprevir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPC3649-206
Record Dates: First submitted 2012-07-04; First posted 2012-07-20 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis C; Chronic Hepatitis C
Keywords: Antisense; miR-122 antagonist; Safety in healthy volunteers; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — miravirsen; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miravirsen sodium (Experimental)
  Interventions: Drug: Miravirsen sodium
- Telaprevir (Active Comparator)
  Interventions: Drug: Telaprevir

INTERVENTIONS:
Drug: Miravirsen sodium — Miravirsen 7 mg/kg to be administered as single subcutaneous injections for a total of 5 doses over a 5 week treatment period.
  Other Names: Miravirsen; SPC3649
  Arms: Miravirsen sodium
Drug: Telaprevir — Telaprevir 750 mg to be administered as single and multiple oral doses over two 7 day treatment periods.
  Other Names: Incivek
  Arms: Telaprevir

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and affect on blood levels of miravirsen and telaprevir when administered together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Weight ≤ 85 kg
* Females of non-childbearing potential (postmenopausal or surgically sterile) or males who are surgically sterile or using an acceptable form of birth control

Exclusion Criteria:

* Current, clinically significant illness or medical condition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The effect of miravirsen on telaprevir pharmacokinetics as determined by AUC0-24h, Cmax and tmax. | Up to 24 hours after dosing.
Safety and tolerability of co-administered miravirsen and telaprevir. | 12 weeks
  Safety and tolerability will be assessed by evaluation of adverse events, physical examinations, vital signs, clinical safety laboratory assessments and electrocardiograms.

SECONDARY OUTCOMES:
The effect of telaprevir on miravirsen pharmacokinetics as determined by AUC0-24h, Cmax and tmax. | Up to 24 hours after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rice, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States